CLINICAL TRIAL: NCT02121197
Title: A Collaborative Retrospective Trial on the Efficacy and Safety of Intravitreal Dexamethasone Implant (Ozurdex) in Patients With Diabetic Macular Edema (DME). THE EUROPEAN DME REGISTRAR STUDY (ARTES)
Brief Title: Retrospective Trial on the Efficacy and Safety of Intravitreal Ozurdex in Patients With Diabetic Macular Edema.
Acronym: ARTES
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Collaborators: European Vision Institute Clinical Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: ECR-RET-2014-07
Record Dates: First submitted 2014-04-22; First posted 2014-04-23 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Diabetic Macular Edema
Keywords: Macular Diabetic Edema; Ozurdex; Retrospective; European; Intra-vitreal injections
MeSH Terms: interventions — Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ozurdex
  Other Names: Dexamethasone

SUMMARY:
To review the safety and efficacy of injections with Ozurdex (700 μg dexamethasone) in clinical practice management of patients with DME.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with diabetes
* DME in the study eye (if both eyes have DME both eyes will be included in analysis)
* BCVA minimum of 20/200 (35 letters)
* Central Macular Thickness (CMT) ≥300 µm
* Patients with DME who were treated with Ozurdex at least twice (baseline is before the first Ozurdex injection).
* Follow up of at least 6 months after the last Ozurdex injection given
* Complete records including BCVA (OCT and Fluorescein Angiography (FA) if available) throughout the follow up

Exclusion Criteria:

* Patients with ME not secondary to Diabetes Mellitus (DM).
* Presence of other retinopathies (AMD, RVO) or visually significant ocular morbidity (e.g. advanced glaucoma, corneal opacity)
* Previous ocular trauma or surgery other than cataract extraction
* Intravitreal triamcinolone ≤6 months before baseline
* Intravitreal bevacizumab, ranibizumab, or pegaptanib <1 months before baseline
* Marked intraocular pressure (IOP) elevation in response to any previous steroid treatment
* Ocular Hypertension (OHT) in the study eye(s)
* IOP >23 mm Hg without antiglaucoma medication
* IOP >21 mm Hg with one antiglaucoma medication
* Use of 2 or more antiglaucoma medications
* Glaucoma - Visual Fields (VF) defect > 4 dB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300-400 patients who have received at least 2 Ozurdex injections for the treatment of DME, were followed for at least 6 months after the last injection and with a minimal BCVA of 20/200 at baseline (before Ozurdex treatment).
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with Best Corrected Visual Acuity (BCVA) from baseline to 4 - 6 months after last injection, with comparison between early (<9 month duration of DME) vs late (≥9 month duration of DME), and naïve vs previously treated patients. | 6 month
  Percentage of patients with Best Corrected Visual Acuity (BCVA) from baseline to 4 - 6 months after last injection, with comparison between early (<9 month duration of DME) vs late (≥9 month duration of DME), and naïve vs previously treated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Anat Loewenstein, Professor, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (25):
- Department of Ophthalmology, Kuopio University Hospital, Kuopio, Finland
- France (5):
  - Department of Ophthalmology, Centre Hospitalier Henri Duffaut,, Avignon
  - Department of Ophthalmology, Croix Rousse University Hospital, Lyon
  - Clinical Trial Unit, Department of Ophthalmology, CHU Nord, Aix Marseille University, Marseille
  - Coscas Eye Clinic, Paris
  - Department of Ophthalmology Lariboisière Hospital, Paris
- Israel (2):
  - Ophthalmology Department, Kaplan Medical Center, Rehovot
  - Department of Ophthalmology Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (6):
  - Ophthalmic Research Unit, Department of Basic Medical Sciences, Neuroscience and Sense Organs, Bari
  - Excellence Eye Research Centre University G. d'Annunzio of Chieti-Pescara, Chieti
  - Department of Ophthalmology University Vita Salute - Scientific Institute of San Raffael, Milan
  - Centre for Clinical Trials, Department of Ophthalmology University of Padova, Padua
  - G.B.Bietti Eye Foundation - IRCCS, Rome
  - Department of Ophthalmology University of Udine, Udine
- Portugal (2):
  - Center for Clinical Trials - Association for Innovation and Biomedical Research on Light and Image, Coimbra
  - Instituto de Retina e Diabetes Ocular de Lisboa (IRL), Lisbon
- Spain (6):
  - Ophthalmology Department, Dos de Maig Hospital, Barcelona
  - Hospital Vall d'Hebrón Department of Ophthalmology, Barcelona
  - Instituto de Microcirugia Ocular, Barcelona
  - Vallés Oftalmologia Research, Barcelona
  - Ophthalmology Department, Hospital de LaPaz, Madrid
  - Servicio de Oftalmologia, Hospital Universitario Y Politecnico de la Fe, Valencia
- Retinal Clinic, St Eriks Hospital, Stockholm, Sweden
- United Kingdom (2):
  - Ophthalmology Clinical Trials Unit Frimley Park Hospital Foundation Trust, Frimley
  - NIHR Moorfields Clinical Research Facility, Moorfields Eye Hospital, NHS Foundation Trust, London